CLINICAL TRIAL: NCT04714710
Title: Evaluation of the Hemodynamic Tolerance of Potassium Canrenoate in Brain-dead Organ Donors: Randomized Controlled Clinical Trial
Brief Title: Potassium Canrenoate in Brain-dead Organ Donors: Randomized Controlled Clinical Trial
Acronym: CANREO-PMO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Study Chair, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-003285-40; 2024-513809-31-00 (EU CTIS Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Brain-dead Organ Donors
Keywords: brain-dead organ donors; mineralocorticoid receptor; Kidney
MeSH Terms: interventions — Canrenoic Acid; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single center, double blinded randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: placebo (sodium chloride solution 0.9%) similar to potassium canrenoate diluted in sodium chloride solution 0.9%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium canrenoate (Experimental): Potassium canrenoate 200mg diluted in SODIUM CHLORIDE SOLUTION 0.9%
  Interventions: Drug: IV Potassium Canrenoate
- Placebo (SODIUM CHLORIDE SOLUTION 0.9%) (Placebo Comparator): SODIUM CHLORIDE SOLUTION 0.9%
  Interventions: Drug: IV Sodium Chloride 0.9 %

INTERVENTIONS:
Drug: IV Potassium Canrenoate — Administration of 200 mg of IV potassium canrenoate (diluted in sodium chloride 0.9%) in brain-dead donors within 10 hours after the diagnosis of brain death and before the departure to the operating room.
  Second administration of potassium canrenoate 6 hours after first administration if the patient is not YET admitted IN the operating room
  Other Names: Drug
  Arms: Potassium canrenoate
Drug: IV Sodium Chloride 0.9 % — Administration of IV sodium chloride 0.9% (placebo) in brain-dead donors within 10 hours after the diagnosis of brain death is made and before the departure to the operating room.
  Second administration of IV sodium chloride 0.9% (placebo) 6 hours after first administration if the patient is not YET admitted IN the operating room.
  Other Names: Placebo
  Arms: Placebo (SODIUM CHLORIDE SOLUTION 0.9%)

SUMMARY:
Given the current organ shortage, improving the quality/efficacy of harvested grafts from expanded criteria donors is essential to substantially increase the number of potential donors. Preclinical studies have shown that blocking the vascular mineralocorticoid receptor (MR) mitigates ischemia-reperfusion injury (I/R) and prevents renal dysfunction following acute kidney injury. Potassium canrenoate is an intravenous MR antagonist. Blocking the MR upstream from aortic cross clamping is likely the most effective strategy to limit I/R injury.

Yet, brain-dead donors are prone to severe hemodynamic instability and polyuria. Consequently, this study seeks to assess the hemodynamic tolerance of the use of potassium canrenoate in this context, as a first step to a large-scale clinical trial testing the impact of this therapeutic intervention on the survival of kidney grafts.

DETAILED DESCRIPTION:
In this single-center, double-blind, placebo-controlled clinical trial, we seek to evaluate the effect of the administration of 200 mg of IV potassium canrenoate vs placebo in brain-dead donors aged 18 years or more - within 10 hours after the diagnosis of brain death is made and before the departure to operating room.

The primary objective is to assess the impact of potassium canrenoate administration vs. placebo on the hemodynamics of brain-dead subjects who are candidates for kidney or multiple organ harvesting (including renal).

The vital status and renal function of kidney recipients will be followed at 3 months, 1 year, 3 years and 10 years from transplant (main secondary objectives)

ELIGIBILITY:
Inclusion Criteria:

* Men, women aged 18 years or older,
* Encephalic death diagnosed either by 2 flat and areactive 30-minute electroencephalograms performed 4 hours apart or by a cerebral angioTDM objectifying a total cessation of intracranial circulation,
* And from whom a removal of one or both kidneys is envisaged (within 6 hours or more), according to the procedures currently in force at the Agence de la Biomédecine,
* Dosage of vasopressor agent amines that have not varied by more than 1 mg/h in the hour preceding inclusion and dose of vasopressor less than 7 mg / h at inclusion,
* euvolemic donor patient at inclusion,
* Benefiting from a Social Security affiliation scheme.
* Signature of consent by a family member or the support person.

Exclusion Criteria:

* Patient having received potassium canrenoate in the 48 hours preceding inclusion in the study,
* Patient on long-term mineralocorticoid receptor antagonist (eplerenone or spironolactone),
* Having a serum potassium concentration> 5.5 mmol / L on inclusion,
* Contraindications to multi-organ removal (infectious, neoplastic causes, etc.),
* Refusal of organ removal expressed by the patient (national register of refusals or reported by the family),
* Probable inability to remove the kidneys: history of urine-renal disease, pre-existing chronic renal failure, morphological abnormalities of the kidneys, renal trauma,
* Patients enrolled in another interventional drug trial,
* Person with a contraindication to potassium canrenoate and/or trometamol,
* Severe renal failure,
* Severe atrioventricular conduction disorders,
* Terminal stage of hepatocellular failure,
* Pregnant, parturient or lactating woman,
* Persons deprived of their liberty by a judicial or administrative decision,
* Minors (non emancipated)
* Adults subject to legal protection measures (guardianship, curatorship, safeguard of justice).
* Person undergoing psychiatric care under articles L3212-1 and L3213-1 of the french Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2033-12-06 (Estimated)

PRIMARY OUTCOMES:
Donor death (cardio circulatory arrest) | from the randomization until the organ removal, up to 24 hours
  The primary endpoint will be a hierarchical composite of events, as described by Felker in 2010 (Circ HF - PMID 20841546) including in descending order:
  A. death (cardio circulatory arrest) before organ removal, B. the inability to perform the renal swab, C. the average hourly dose of noradrenaline / adrenaline between randomization and departure to the operating room, D. the average hourly volume of crystalloids and / or colloids used between randomization and departure to the operating room.
Inability to perform kidney harvest | Up to 24 hours, in the organ removal during surgery
  The primary endpoint will be a hierarchical composite of events, as described by Felker in 2010 (Circ HF - PMID 20841546) including in descending order:
  A. death (cardio circulatory arrest) before organ removal, B. the inability to perform the renal swab, C. the average hourly dose of noradrenaline / adrenaline between randomization and departure to the operating room, D. the average hourly volume of crystalloids and / or colloids used between randomization and departure to the operating room.
The average hourly dose of norepinephrine or epinephrine | From the randomization until the departure to the operating room, up to 24 hours
  The primary endpoint will be a hierarchical composite of events, as described by Felker in 2010 (Circ HF - PMID 20841546) including in descending order:
  A. death (cardio circulatory arrest) before organ removal, B. the inability to perform the renal swab, C. the average hourly dose of noradrenaline / adrenaline between randomization and departure to the operating room, D. the average hourly volume of crystalloids and / or colloids used between randomization and departure to the operating room.
The average hourly volume of crystalloids and / or colloids | from the randomization until the departure to the operating room, up to 24 hours
  The primary endpoint will be a hierarchical composite of events, as described by Felker in 2010 (Circ HF - PMID 20841546) including in descending order:
  A. death (cardio circulatory arrest) before organ removal, B. the inability to perform the renal swab, C. the average hourly dose of noradrenaline / adrenaline between randomization and departure to the operating room, D. the average hourly volume of crystalloids and / or colloids used between randomization and departure to the operating room.

SECONDARY OUTCOMES:
Mortality rate of the kidney recipients | 3 months, 1 year, 3 years, and 10 years from kidney transplant
  The number of patients dead after kidney transplantation
Serum creatinine (in μmol / L) of kidney recipients | 3 months, 1 year, 3 years, and 10 years from kidney transplant
  With estimation of the glomerular filtration rate (GFR) according to CKD-EPI (in mL / min / 1.73m2).
Percentage of kidney recipients dependent on dialysis and / or with an estimated GFR <20 mL / min / 1.73m² | 3 months after kidney transplant
  Number of patients on dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GUERCI, MD, PhD, Principal Investigator — CHRU de NANCY; Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY; Patrick ROSSIGNOL, MD-PhD, Study Chair — CHRU de NANCY; Luc FRIMAT, MD-PhD, Study Chair — CHRU de NANCY; Hélène GREGOIRE, MD, Study Chair — CHRU de NANCY
Locations (1):
- CHRU de NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reseanable request to the principal investigator in compliance with french regulations.

REFERENCES:
- [Derived] Belarif L, Girerd S, Jaisser F, Lepage X, Merckle L, Duarte K, Girerd N, Guerci P. Potassium canrenoate in brain-dead organ donors: a randomised controlled clinical trial protocol (CANREO-PMO). BMJ Open. 2023 Oct 11;13(10):e073831. doi: 10.1136/bmjopen-2023-073831. PMID 37821131

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04714710/SAP_001.pdf